CLINICAL TRIAL: NCT04872335
Title: Comparative Effects of Gong's Mobilization With Gradually Graded Exercise Therapy for Chronic Neck Pain Among the Electronic Gadgets Users.
Brief Title: Comparative Effects of Gong's Mobilization With Gradually Graded Exercise Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Rabiya Noor, Associate Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0104
Record Dates: First submitted 2021-03-26; First posted 2021-05-04 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain; Neck Pain; Shoulder Syndrome
Keywords: Gong's Mobilization; Gradually graded exercise therapy
MeSH Terms: conditions — Chronic Pain; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong's Mobilization (Experimental): Subjects received gong's mobilization three times in a week for 4 weeks.
  Interventions: Other: Gong's Mobilization
- Gradually Graded Exercise Therapy (Experimental): Subjects received gradually graded exercise therapy three times in a week for 4 weeks.
  Interventions: Other: Gradually Graded Exercise Therapy

INTERVENTIONS:
Other: Gong's Mobilization — Group A received Gong's mobilization and common treatnent (TENs,Hot pack and cervical stretches). Gong's mobilization which is concurrent application of Apophyseal joint gliding and end range passive physiological movements while the subject's cervical postures are passively Neutral in order to induce Normal Cervical Extension. The Subjects in Group A were treated three times in a week for 4 weeks.
  Arms: Gong's Mobilization
Other: Gradually Graded Exercise Therapy — The Subjects in Group B were received Exercise Therapy and common treatment (TENs, Hot pack and cervical stretches) three times in a week continue for 4 weeks . Each exercise session will take 30 min. It will be consisted of 5 min warm-up exercises, 20 min stabilization exercises, 5 min cool-down, and stretching exercises including neck and shoulder girdle muscles.
  The aim of Exercise program was to create a neutral spine and activate deep muscles of the cervical spine. The patients were educated to maintain neutral spine during the exercises and throughout the day as much as possible.
  Scapulothoracic stabilization exercises were included_ specific exercises for the muscles affecting scapular orientation related to neck pain. The subjects were educated to maintain the positions and contractions during the exercises including scapular retraction, eccentric scapular retraction, and combined scapular retraction with shoulder lateral rotation, forward punch, and dynamic hug.
  Arms: Gradually Graded Exercise Therapy

SUMMARY:
This project was a Randomized clinical trial conducted to find out the Comparative Effects of Gong's Mobilization with Gradually Graded Exercise Therapy for Chronic Neck Pain among the users of Electronic Gadgets so that we can have best treatment option for patients.

DETAILED DESCRIPTION:
The study design was a Randomized Clinical Trial. For the study data was collected from sports and spine professionals. Sample size was calculated with the help of Epitool calculator. The study will be completed in 6 months duration. Neck Disability Index (NDI), Numeric Pain Rating Scale (NPRS) for pain intensity and Universal Goniometers for measuring (ROMs) and Forward head posture (FHP) were assessed before and 4 weeks after the treatment through the craniovertebral angle (CVA) measured from a digitized, lateral-view photograph of each subject. All the subjects were selected using Non Probability convenient sampling technique. The Subjects were randomly assigned to one of the following two groups: Gong's Mobilization (Group 1) or Gradually Graded Exercise Therapy (Group 2).This study was conducted in accordance with the rules of the Declaration of Helsinki. Written Informed consent were taken from all the subjects before participating in this trial. SPSS 25 was used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:• Subjects with an age range of 15 to 65 years having Chronic neck pain for more than 3 months and subjects having a baseline NDI score of atleast 20% (10 points).

-

Exclusion Criteria:

* • Cervical stenosis

  * History of traumatic Injury
  * Previous surgery related to cervical spine
  * Hypermobility
  * Cancer
  * Inflammatory rheumatologic diseases
  * Severe psychological disorders
  * Being pregnant and
  * Intervention including exercise or physical therapy in the last 3 months.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity by 'Numeric Pain Rating Scale' | Baseline (pre treatment readings), Immediate after treatment and post treatment readings( at 4th week)
  Change in pain from baseline was measured at 12th session. The Numerical Pain Rating Scale (NPRS) is an 11 point pain scale that is completed by subject himself, under the supervision of researcher.
Change in Neck disability Index 'NDI' score | Baseline (pre treatment readings), Immediate after treatment and post treatment readings( at 4th week)
  Change in Neck disability Index score 'NDI' from baseline was measured at 12th session. This questionnaire or tool has been designed to give us information as to how neck pain of the subject has affected his/her ability to manage in everyday life.

SECONDARY OUTCOMES:
Change in Cervical Range of Motion (ROM) measured by Universal Goniometer. | Baseline (pre treatment readings), Immediate after treatment and post treatment readings( at 4th week)
  Change in Cervical Range of motion (ROM) from baseline was measured at 12th session.
Change in Craniovertebral angle CVA measured from a digitized, lateral-view photograph of each subject. | Baseline (pre treatment readings), Immediate after treatment and post treatment readings( at 4th week)
  Change in Craniovertebral angle (CVA) from baseline was measured at 12th session. Craniovertebral angle (CVA) is a factor that significantly influences pain in those individuals with a forward head posture (FHP). Craniovertebral angle (CVA) (the angle between the horizontal line passing through C7 and a line extending from the tragus of the ear to C7).

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah International University, Lahore, Punjab Province
  - Riphah IU, Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celenay ST, Kaya DO, Akbayrak T. Cervical and scapulothoracic stabilization exercises with and without connective tissue massage for chronic mechanical neck pain: A prospective, randomised controlled trial. Man Ther. 2016 Feb;21:144-50. doi: 10.1016/j.math.2015.07.003. Epub 2015 Jul 15. PMID 26211422
- [Background] Gong W. The effects of cervical joint manipulation, based on passive motion analysis, on cervical lordosis, forward head posture, and cervical ROM in university students with abnormal posture of the cervical spine. J Phys Ther Sci. 2015 May;27(5):1609-11. doi: 10.1589/jpts.27.1609. Epub 2015 May 26. PMID 26157273
- [Background] McLean SM, Klaber Moffett JA, Sharp DM, Gardiner E. A randomised controlled trial comparing graded exercise treatment and usual physiotherapy for patients with non-specific neck pain (the GET UP neck pain trial). Man Ther. 2013 Jun;18(3):199-205. doi: 10.1016/j.math.2012.09.005. Epub 2012 Oct 22. PMID 23085116
- [Background] Kim DH, Kim CJ, Son SM. Neck Pain in Adults with Forward Head Posture: Effects of Craniovertebral Angle and Cervical Range of Motion. Osong Public Health Res Perspect. 2018 Dec;9(6):309-313. doi: 10.24171/j.phrp.2018.9.6.04. PMID 30584494